CLINICAL TRIAL: NCT01435772
Title: A Long-Term Study for Extended BMN 701 Treatment of Patients With Pompe Disease Who Have Participated in a BMN 701 Study
Brief Title: Extension Study for Patients Who Have Participated in a BMN 701 Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated because BioMarin decided to end the overall development program based on competing corporate priorities.
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POM-002; 2011-001805-28 (EudraCT Number)
Record Dates: First submitted 2011-09-08; First posted 2011-09-19 (Estimated); Results first posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Pompe Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMN 701 20mg/kg (Experimental): BMN 701 20mg/kg IV every other week
  Interventions: Biological: BMN 701
- BMN 701 10mg/kg (Experimental): BMN 701 10mg/kg IV every other week
  Interventions: Biological: BMN 701
- BMN 701 5mg/kg (Experimental): BMN 701 5mg/kg IV every other week
  Interventions: Biological: BMN 701

INTERVENTIONS:
Biological: BMN 701 — GILT-tagged recombinant human GAA

SUMMARY:
This is a Phase 2 open-label, multiple dose study of BMN 701 administered by IV infusion every 2 weeks (qow) to patients with late-onset Pompe disease.

ELIGIBILITY:
Inclusion Criteria:

* Have completed a prior BMN 701 clinical development study;
* Have provided written informed consent after the nature of the study has been explained prior to performance of any study-related procedures. Minors may participate as long as they provide written assent after the nature of the study has been explained to them and after their parent, or legal guardian has provided written informed consent, prior to the performance of any study-related procedures;
* Have been diagnosed with late-onset Pompe Disease, based on the entry criteria of a prior BMN 701 study;
* If sexually active, be willing to use 2 known effective methods of contraception from Screening until 4 months after the last dose of study-drug;
* If female, and not considered to be of childbearing potential, be at least 2 years post-menopausal, or have had tubal ligation at least 1 year prior to screening, or have had a total hysterectomy;
* If female, and of childbearing potential, have a negative pregnancy test during the Screening Period and at the Baseline visit, and be willing to have additional pregnancy tests during the study;
* Have the ability to comply with the protocol requirements, in the opinion of the Investigator.

Exclusion Criteria:

* Have received any experimental or approved therapy for Pompe disease, other than BMN 701, subsequent to completion of a BMN 701 study and prior to entry into POM-002;
* Have received, or are anticipated to receive, any investigational medication, other than BMN 701, within 30 days prior to the first dose of study-drug;
* Are breastfeeding at screening or planning to become pregnant (self or partner) at any time during the study;
* Have a medical condition or extenuating circumstance that, in the opinion of the Investigator, might compromise the patient's ability to comply with the protocol requirements or compromise the patient's well being or safety.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2016-09-09 (Actual); Study Completion 2016-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — BioMarin Pharmaceutical
Locations (12):
- United States (4):
  - Univ of California San Diego School of Medicine, San Diego, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, North Adelaide, South Australia
- Hôpital Pitié-Salpêtrière, Paris, France
- Villa Metabolica, ZKJM MC University Mainz, Mainz, Germany
- Auckland City and Starship Children's Hospital, Auckland, New Zealand
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Free Hospital, London
  - Salford Royal NHS Foundation Trust, Salford

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN 701 5 mg/kg: IV infusion at dose levels of 5 mg/kg
- BMN 701 10 mg/kg: IV infusion at dose levels of 10 mg/kg
- BMN 701 20 mg/kg: IV infusion at dose levels of 20 mg/kg
Period: Overall Study
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Started | 3 | 3 | 15
Completed | 0 | 0 | 0
Not Completed | 3 | 3 | 15
Not completed — Adverse Event | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 3
Not completed — Other - study termination | 2 | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 15 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (6.66) | 42.7 (13.05) | 50.1 (5.28) | 49.4 (7.03)
Age, Customized [Count of Participants; unit: Participants]
  18-65 years | 3 | 3 | 15 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 6 | 8
  Male | 3 | 1 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 15 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Black or African American | 0 | 0 | 0 | 0
  Race: White | 3 | 3 | 14 | 20
  Race: Other | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 1 | 1 | 4 | 6
  France | 0 | 0 | 1 | 1
  Germany | 0 | 0 | 1 | 1
  United Kingdom | 0 | 0 | 6 | 6
  United States | 2 | 2 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive Anti-BMN 701 Antibody
Description: Status of Anti-BMN 701 antibody is corresponding to the test results of blood samples.
Time Frame: Baseline, Week 144
Population: Full Analysis Set. Please note the overall number of participants reflects the number of patients in that arm, while the outcome measurement number of participants reflects the number of patients for which data is available and analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Participants
  Baseline: number analyzed (Participants) | 2 | 1 | 12
  Baseline | 2 | 1 | 11
  Week 144: number analyzed (Participants) | 2 | 2 | 10
  Week 144 | 2 | 2 | 10

2. Primary Outcome: Number of Participants With a Positive Anti-BMN 701 Antibody Response
Description: Status of Anti-IGF-I antibody is corresponding to the test results of blood samples
Time Frame: Baseline, Week 144
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Participants
  Baseline | 0 | 2 | 0
  Week 144: number analyzed (Participants) | 2 | 2 | 10
  Week 144 | 0 | 1 | 5

3. Primary Outcome: Number of Participants With a Positive Anti-BMN 701 Antibody Response
Description: Status of Anti-IGF-II antibody is corresponding to the test results of blood samples
Time Frame: Baseline, Week 144
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Participants
  Baseline | 1 | 2 | 2
  Week 144: number analyzed (Participants) | 2 | 2 | 10
  Week 144 | 0 | 2 | 7

4. Secondary Outcome: Percent Predicted Maximal Inspiratory Pressure (MIP)
Description: Pulmonary Function Test: Percent Predicted Maximal Inspiratory Pressure
Time Frame: Baseline, Week 144
Population: Full Analysis Set. No data collected for outcomes with 0 participants analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Predicted
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 0 | 3 | 15
Percent of Predicted
  Baseline |  | 39.53 (21.868) | 40.2 (25.863)
  Change from Baseline to Week 144: number analyzed (Participants) | 0 | 2 | 11
  Change from Baseline to Week 144 |  | 21.17 (14.537) | 18.48 (18.599)

5. Secondary Outcome: Percent Predicted Maximum Expiratory Pressure (MEP)
Description: Pulmonary Function Test: Percent Predicted Maximum Expiratory Pressure
Time Frame: Baseline, Week 144
Population: Full Analysis Set. No data collected for outcomes with 0 participants analyzed.
Measure: Mean (Standard Deviation); unit: Percent of Predicted
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 0 | 3 | 15
Percent of Predicted
  Baseline |  | 31.07 (6.641) | 36.7 (15.939)
  Change from Baseline to Week 144: number analyzed (Participants) | 0 | 2 | 11
  Change from Baseline to Week 144 |  | -0.28 (5.841) | 5.11 (16.395)

6. Secondary Outcome: 6 Minutes Walk Test (Meters)
Description: Distance walked within 6 minutes
Time Frame: Baseline, Week 144
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
meter
  Baseline | 334 (227.119) | 360 (51.403) | 363.8 (157.818)
  Change from Baseline to Week 144: number analyzed (Participants) | 3 | 2 | 11
  Change from Baseline to Week 144 | -36 (90.508) | -120.75 (67.529) | 9.5 (77.572)

7. Secondary Outcome: Maximum Voluntary Ventilation (MVV)
Description: Pulmonary function test: Maximum Voluntary Ventilation (MVV)
Time Frame: Baseline, Week 144
Population: Full Analysis Set. No data collected for outcomes with 0 participants analyzed.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 0 | 3 | 15
L/min
  Baseline |  | 76 (41.037) | 68.08 (26.74)
  Change from Baseline to Week 144: number analyzed (Participants) | 0 | 2 | 11
  Change from Baseline to Week 144 |  | 13.5 (13.435) | 2.24 (11.635)

8. Secondary Outcome: Percent Predicted Upright Forced Vital Capacity (FVC)
Description: Pulmonary function test: Percent Predicted Upright Forced Vital Capacity
Time Frame: Baseline, Week 144
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Percent Predicted
  Baseline | 69.33 (19.732) | 67.33 (26.577) | 57.13 (18.677)
  Change from Baseline to Week 144: number analyzed (Participants) | 3 | 2 | 11
  Change from Baseline to Week 144 | -8.33 (7.095) | -0.5 (4.95) | -2 (8)

9. Secondary Outcome: Percent Predicted Upright Forced Vital Capacity (FVC)
Description: Pulmonary function test: Percent Predicted Upright Forced Vital capacity
Time Frame: Baseline, Week 144
Population: Full Analysis Set.
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
Percent Predicted
  Baseline: number analyzed (Participants) | 3 | 3 | 12
  Baseline | 36.67 (17.954) | 47.67 (32.578) | 44.25 (21.55)
  Change from Baseline to Week 144: number analyzed (Participants) | 3 | 2 | 7
  Change from Baseline to Week 144 | -4.33 (9.452) | 4.5 (26.163) | -3.43 (6.901)

10. Secondary Outcome: Change From Baseline in Urine Tetrasaccharide Concentration at Week 144
Description: Change from Baseline in Urine Tetrasaccharide Concentration at Week 144
Time Frame: Baseline, Week 144
Population: Full Analysis Set. No data collected for outcomes with 0 participants analyzed.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 0 | 2 | 10
mmol/mol |  | -0.2 (3.394) | -1.07 (0.975)

11. Secondary Outcome: Plasma IGF-I Concentration
Description: Plasma IGF-I concentration from lab
Time Frame: Baseline, Week 144
Population: Full Analysis Set. No data collected for outcomes with 0 participants analyzed. Please note: the overall number of participants reflects the number of patients in that arm, while the outcome measurement number of participants reflects the number of patients for which data is available and analyzed.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 2 | 2 | 15
nmol/L
  Baseline: number analyzed (Participants) | 0 | 0 | 11
  Baseline |  |  | 20.26 (6.465)
  Week 144: number analyzed (Participants) | 2 | 2 | 11
  Week 144 | 26.98 (1.379) | 18.4 (7.078) | 17.62 (5.878)

12. Secondary Outcome: Plasma IGF-II Concentration
Description: Plasma IGF-II concentration from lab
Time Frame: Baseline, Week 144
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 3 | 15
nmol/L
  Baseline: number analyzed (Participants) | 0 | 1 | 6
  Baseline |  | 702 (0) | 496.83 (113.417)
  Week 144: number analyzed (Participants) | 3 | 2 | 11
  Week 144 | 467.67 (117.142) | 559.5 (140.714) | 698.82 (228.948)

13. Secondary Outcome: Insulin-like Growth Factor Binding Protein 3 (IGFBP3)
Description: insulin-like growth factor binding protein 3 from lab
Time Frame: Baseline, Week 144
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg
Number analyzed (Participants) | 3 | 2 | 15
nmol/L
  Baseline: number analyzed (Participants) | 0 | 0 | 11
  Baseline |  |  | 150.45 (23.914)
  Week 144: number analyzed (Participants) | 3 | 2 | 11
  Week 144 | 157.33 (41.477) | 209 (39.598) | 146.64 (33.587)

ADVERSE EVENTS:
Time Frame: 284.9 weeks (maximum exposure) +4 weeks follow up
Groups:
- BMN 701 5 mg/kg: BMN 701 5 mg/kg
- BMN 701 10 mg/kg: BMN 701 10 mg/kg
- BMN 701 20 mg/kg: BMN 701 20 mg/kg
- Total: Total
Arm/Group | BMN 701 5 mg/kg | BMN 701 10 mg/kg | BMN 701 20 mg/kg | Total
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 7/15 | 10/21
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 15/15 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 701 5 mg/kg (N=3) | BMN 701 10 mg/kg (N=3) | BMN 701 20 mg/kg (N=15) | Total (N=21)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaphylactoid reaction (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 701 5 mg/kg (N=3) | BMN 701 10 mg/kg (N=3) | BMN 701 20 mg/kg (N=15) | Total (N=21)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 5 (49) | 7 (51)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Androgen deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blindness transient (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (3) | 3 (5)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (5) | 5 (7)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 7 (13) | 7 (13)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (29) | 8 (31)
Painful defaecation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (5) | 1 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Application site erythema (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 5 (19) | 6 (20)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (18) | 0 (0) | 8 (16) | 10 (34)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 2 (10) | 3 (11)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 3 (7) | 4 (8)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Infusion site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Infusion site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 4 (5) | 5 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 3 (8) | 3 (8)
Pain (General disorders) | 2 (2) | 0 (0) | 1 (2) | 3 (4)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Blister infected (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 4 (9) | 6 (11)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 4 (7) | 5 (8)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (3) | 2 (6) | 7 (11) | 10 (20)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 2 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (5) | 1 (1) | 6 (9) | 9 (15)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (22) | 2 (5) | 7 (26) | 12 (53)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 2 (2) | 3 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (5) | 1 (1) | 1 (1) | 4 (7)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ammonia increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 7 (14) | 7 (14)
Blood immunoglobulin E increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Complement factor increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary physical examination abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tryptase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (19) | 1 (30) | 14 (106) | 16 (155)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (8) | 1 (1) | 7 (18) | 10 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1) | 7 (10) | 11 (17)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (9) | 4 (10)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (4)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 8 (14) | 10 (16)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 1 (5) | 8 (11) | 10 (17)
Headache (Nervous system disorders) | 2 (7) | 1 (4) | 9 (30) | 12 (41)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tunnel vision (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1) | 2 (2) | 4 (5)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (4) | 1 (1) | 4 (6) | 6 (11)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Sleep terror (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (8) | 3 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 9 (26) | 10 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 5 (12) | 7 (15)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (40) | 1 (40)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (4)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 1 (4)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 3 (4) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (14) | 4 (14)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (3) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (5) | 1 (1) | 4 (7)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (3)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (8) | 1 (1) | 2 (3) | 6 (12)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 4 (8) | 4 (8)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hot flush (Vascular disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (6)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (6)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (6) | 3 (6)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes